CLINICAL TRIAL: NCT03146130
Title: Study of the Efficacy of N-acetylcysteine (NAC) on Impulse Control Disorders (TCI) Induced by Dopaminergic Treatments in Parkinson's Disease
Brief Title: Study of the Efficacy of N-acetylcysteine (NAC) on Impulse Control Disorders
Acronym: NoISE-PD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI2016_843_0002
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Impulse Control Disorder; Parkinson
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient treated with N-acetylcysteine (Active Comparator): Patients randomise in the drug group
  Interventions: Biological: Variation of behaviors of Parkinson's disease
- Patient treated with placebo (Placebo Comparator): Patients randomise in the placebo group
  Interventions: Biological: Variation of behaviors of Parkinson's disease

INTERVENTIONS:
Biological: Variation of behaviors of Parkinson's disease — Variation of hyper dopaminergic behaviors of Parkinson's disease

SUMMARY:
Impulse control disorders encountered in Parkinson's disease (PD) are induced by dopaminergic medications and their frequency is estimated to be nearly 20%, mainly under dopaminergic agonists (AD).

DETAILED DESCRIPTION:
Impulse control disorders encountered in Parkinson's disease (PD) are induced by dopaminergic medications and their frequency is estimated to be nearly 20%, mainly under dopaminergic agonists (AD). They constitute a major public health issue due to their sometimes dramatic socio-occupational and judicial consequences. Most often the therapeutic strategy is to reduce or even stop AD, which can lead to withdrawal symptoms, apathy or aggravation of motor signs.

N-acetylcysteine (NAC) may have an interest in the treatment of ICD. This molecule reduces "craving" in addictions by substance abuse, but also in behavioral addictions, with as a potential mechanism a reduction in levels of plasma alphasynuclein.

The main objective of this randomized, double-blind, placebo-controlled, multicenter controlled trial is to demonstrate that a 10-week NAC add-on treatment, compared to placebo, improves the behavioral addictions of Moderate in the MP. The main endpoint will be the variation of the subdivision of the hyperdopaminergic behaviors of the Ardouin Parkinson's Disease Behavioral Assessment (ECMP) scale between the baseline and after 10 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to UKPDSBB criteria
* Subject aged 18 to 80
* Presence of a mild to moderate impulse control disorder defined by an ECD hyperdopaminergic sub-score (part IV) between 3 and 22 associated with the investigator's assessment
* MMSE ≥ 24
* Ongoing treatment with dopaminergic agonist and / or levodopa
* No change in antiparkinsonian and / or psychotropic treatment in the month preceding inclusion
* Expected stability of antiparkinsonian and / or psychotropic treatment during the study period
* Informed patient consent
* Patient supported by social security
* Presence of a caregiver

Exclusion Criteria:

* Severe TCI defined by a hyperdopaminergic sub-score at ECMP (part IV) greater than 23 associated with the investigator's assessment
* Patient with TCI suspected of having serious legal and / or relationship problems during the study period
* Adaptation of the anti-parkinsonian and / or psychotropic treatment (cf section 6.2) probably necessary during the duration of the study
* Patient treated with naltrexone, amantadine, antipsychotic in the 6 weeks prior to inclusion
* Patient under tutorship or curatorship
* History of hypersensitivity to any of the components or to any of the excipients
* Fructose intolerance, glucose-galactose malabsorption syndrome or sucrase / isomaltase deficiency
* Gastrointestinal duodenal ulcer in progress
* Pregnancy, breastfeeding
* Patients with contra-indicated treatments in association with NAC
* Patient with phenylketonuria
* Patients with proven difficulty in expectorating
* Patients with an asthmatic risk that can lead to bronchospasm
* Patients with intolerance to histamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the variation of the scale of the behavioral evaluation | 11 weeks
  show that a 10-week treatment with N-acetylcysteine compared to placebo improves the mild-to-moderate impulse control disorders induced by dopaminergic medications in Parkinson's disease.
  The primary endpoint is the change in score from Part IV of the Ardouin Parkinson's Behavioral Assessment of Parkinson's Disease (ECMP) (ECMP IV), which evaluates hyperdopaminergic behaviors between the baseline and after 10 weeks. treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa TIR, Dr, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France